CLINICAL TRIAL: NCT02476877
Title: A Pilot, Proof-of-concept Cohort Study of the Prevalence of Comorbid Mental Illness and Substance Abuse
Status: Completed | Type: Observational
Sponsor: Advanced Clinical Laboratory Solutions, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ACLS-COMORBIDITY-001
Record Dates: First submitted 2015-06-16; First posted 2015-06-22 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Schizophrenia; Drug Abuse; Anxiety Disorder; Bipolar Disorder; Major Depression
Keywords: comorbidity; epidemiology; mental illness; drug abuse
MeSH Terms: conditions — Schizophrenia; Substance-Related Disorders; Anxiety Disorders; Bipolar Disorder; Depressive Disorder, Major; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Each subject will be asked to provide a urine sample (minimum of 5 mL). If a subject cannot provide a urine sample, a sample of oral fluids (1 mL) will be obtained.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Prescribed-drug treatment group: Eight hundred (800) subjects of which 200 subjects in each of the four mental illnesses will continue to receive prescription drug therapy (as prescribed by their physician/psychiatrist) and counseling to treat their mental illness.
- Naïve drug group: Two hundred (200) subjects of which about 50 subjects in each of the four mental illnesses will be initially drug naïve (i.e. currently not taking psychotropic drugs) at the beginning of the study and continue to be drug naïve until the end of the study (6 months) as they receive counseling for their mental illness.

SUMMARY:
The prevalence estimates for specific mental disorders and illicit drugs have been separately reported in U.S. government surveys. Less is known about the rates for specific comorbid conditions, e.g., schizophrenia and substance abuse, major depression and substance abuse, bipolar disorder and substance abuse, and anxiety disorder and substance abuse. The effects that different demographic characteristics (ethnic background, family medical history, age, living conditions [e.g., living with a single parent]) have on the prevalence of comorbid mental illness and substance abuse also have not been considered. More should be known about the duration of substance abuse in different mental illnesses among those undergoing treatment, and whether specific types of drugs are associated with specific mental illnesses.

In this study, Advanced Clinical Laboratory Solutions, Inc. will investigate the prevalence rates for the specific comorbid conditions and demographic relationships described above. This multi-site, proof-of-concept cohort study will analyze urine or oral fluid samples from 1,000 subjects diagnosed with one of four mental illnesses (schizophrenia, major depression, bipolar disorder, or anxiety disorder) as determined by DSM-IV (The Fourth Edition of the Diagnostic and Statistical Manual of Mental Disorders). The samples will be analyzed for both prescription drug compliance and illicit substance abuse. Urine or oral fluid samples will be collected at three time points: 1) immediately after enrollment and obtaining informed consent, 2) randomly within 2 to 4 months of the study, and 3) at the end of the study (6 months).

DETAILED DESCRIPTION:
The National Comorbidity Survey Replication (NCS-R), conducted between 2001 and 2003, reported U.S. lifetime prevalence estimates for anxiety disorders (28.8%), mood disorders (20.8%), impulse-control disorders (24.8%), substance use disorders (14.6%), and any disorders (46.4%). Some of these mental conditions start as early as 11 years of age. According to the NCS-R, about half of Americans met or will meet the criteria for a DSM-IV disorder sometime in their life.

The rates for illicit drug use have also been reported. The highest rate of illicit drug use in the U.S. was among 18 to 20 year-olds (23.9%), while the next highest rate occurred among 21-25 year-old adults (19.7%). Males were more likely than females to be users of illicit drugs. As compared to whites (9.2%), rates for illicit drug use were higher among Blacks (11.3%), Native Americans (12.7%) and among persons of two or more ethnic backgrounds (14.8%). Marijuana is the most used drug (18.9 million) followed by pain relievers (6.8 million) and cocaine (1.6 million).

Mental illness surveys have shown that mental disorders are often associated with the risk for substance abuse. The National Survey on Drug Use and Health indicated that, in 2002, approximately 23% (4 million) of adults with serious mental illness were also dependent on or abused alcohol or an illicit drug. However, more than half of the adults (2 million) with co-occurring serious mental illnesses and substance abuse (i.e., comorbidity) received neither mental health nor substance abuse treatment during the previous year.

While the prevalence estimates for specific mental disorders and illicit drugs have been separately reported in U.S. government surveys, less is known about the rates for specific comorbid conditions, e.g., schizophrenia and substance abuse, major depression and substance abuse, bipolar disorder and substance abuse, and anxiety disorder and substance abuse. The effects that different demographic characteristics (ethnic background, family medical history, age, living conditions [e.g., living with a single parent]) have on the prevalence of comorbid mental illness and substance abuse have not been considered in detail. Additionally, more should be known about the duration of substance abuse in different mental illnesses among those undergoing treatment, and whether specific types of drugs are associated with specific mental illnesses.

In this study, Advanced Clinical Laboratory Solutions, Inc. will investigate the prevalence rates for the specific comorbid conditions and demographic relationships described above. This multi-site, proof-of-concept cohort study will analyze urine or oral fluid samples from 1,000 subjects diagnosed with one of four mental illnesses (schizophrenia, major depression, bipolar disorder, or anxiety disorder) as determined by DSM-IV. The samples will be analyzed for both prescription drug compliance and illicit substance abuse. Urine or oral fluid samples will be collected at three time points: 1) immediately after enrollment and obtaining informed consent, 2) randomly within 2 to 4 months of the study, and 3) at the end of the study (6 months).

The results of this study will provide new detailed information about the comorbid relationship between specific mental illnesses and substance abuse. Oral fluid and urinalysis screening will provide compliance information (for drugs prescribed for mental illness treatment) and may reveal illicit drug use by their patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has granted written informed consent.
2. Male or female subject aged 18 years and older.
3. Diagnosed with one of four mental illnesses (schizophrenia, major depression, bipolar disorder, or anxiety disorder) as determined by DSM-IV.
4. Residents of households, non-institutional group quarters (e.g., shelters, rooming houses, and dormitories), and civilians living on military bases.

Exclusion Criteria:

1. Subjects younger than 18 years of age.
2. Subjects who require a legally authorized representative.
3. Subjects who have multiple psychiatric diagnoses.
4. Homeless persons who do not use shelters, military personnel on active duty, residents of jails, and residents of institutional group quarters such as hospitals.
5. Subjects who are not diagnosed with one of four mental illnesses (schizophrenia, major depression, bipolar disorder, or anxiety disorder) as determined by DSM-IV.
6. A medical condition that, in the PI's opinion, could adversely impact the subject's participation or safety, or affect the conduct of the study, or interfere with the urine or oral fluid assessments.
7. Subjects who are terminally ill and/or having an acute/chronic illness such as cancer that will affect their compliance to prescribed medicine.
8. Subject who is not able to understand the nature, importance, or consequences of the study.
9. Subject who has been treated with an investigational drug, device, or therapy within 30 days prior to screening.
10. Subject who has significant or unstable hypertension, vascular disease, or other condition that would interfere with the completion of the study.
11. The subject who has a serious or unstable illness or is not in good general health.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female subjects who are aged 18 years and older with one of four mental illnesses (schizophrenia, major depression, bipolar disorder, or anxiety disorder) as determined by DSM-IV criteria. Subjects who have multiple psychiatric diagnoses will be excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2014-06; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Prevalence of the co-morbidity of mental illness with substance abuse | 1 year
  The primary outcome measure of this study is to determine the prevalence of the co-morbidity of mental illness with substance abuse among a cohort of adults residing in the metropolitan area of New York City. Diagnoses of the four mental illnesses considered in the study (schizophrenia, major depression, bipolar disorder, or anxiety disorder) will be based on DSM-IV criteria. Approximately 1,000 subjects will be enrolled in order to obtain about 3,000 urine or oral fluid samples. Subjects who have multiple psychiatric diagnoses will be excluded from the study.

SECONDARY OUTCOMES:
Association between demographic characteristics and the prevalence of substance abuse in each of the four mental illnesses | 1 year
  A secondary outcome measure is the association between demographic characteristics (ethnic background, family medical history, age, living conditions [e.g., living with a single parent]) and the prevalence of the co-morbidity of mental illness with substance abuse.
Duration of substance abuse in each of the four mental illnesses | 1 year
  A secondary outcome measure is the duration of substance abuse in each of the four mental illnesses.
Types of drugs associated with each of the four mental illnesses | 1 year
  A secondary outcome measure is the types of drugs that are associated with each of the four mental illnesses.

CONTACTS AND LOCATIONS:
Overall Officials: Leonid Reyfman, MD, Principal Investigator — Advanced Clinical Laboratory Solutions, Inc.
Locations (1):
- Advanced Clinical Laboratory Solutions, Inc., Brooklyn, New York, United States